CLINICAL TRIAL: NCT02584686
Title: Intracavernosal Injection of Botulinum Toxin Type A in the Treatment of Vascular Erectile Dysfunction Not Responding to Oral and Intracavernous Therapy
Brief Title: Intracavernosal Injection of Botulinum Toxin Type A in the Treatment of Vascular Erectile Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hussein Ghanem, Professor and Chairman, Department of Andrology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1121015
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Vasculogenic Erectile Dysfunction
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (BTX) A Group (Experimental): The treatment group will be injected intracavernously with a trimix solution for colour Doppler assessment, followed, on a separate day by 50 units of Botulinum toxin (BTX) A.
  Interventions: Drug: Botulinum Toxin Type A
- Saline Group (Placebo Comparator): The control group, 12 patients, will be injected with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) during penile colour Doppler assessment followed on a separate day with a normal saline injection.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — The treatment group will be injected intracavernously with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) for colour Doppler assessment, followed next day by 50 units of BTX-A.
  Arms: (BTX) A Group
Drug: Normal Saline — The control group, 12 patients, will be injected with a trimix solution during penile colour Doppler assessment followed next day with a normal saline injection.
  Arms: Saline Group

SUMMARY:
Evidence has been arising that Botulinum toxin injections can relax smooth muscles fibers in the treatment of obesity and hyperactive bladder. Would a similar effect on cavernosal smooth muscles help in the treatment of resistant erectile dysfunction not responding to medical and injection therapy, thus avoiding surgical treatment options.

The treatment group will be injected intracavernously with 50 units of BTX-A. The control group, 12 patients, will be injected with a normal saline injection.

DETAILED DESCRIPTION:
24 males with will be included in the study. All will be subjected for full history taking, general and genital examination. Penile duplex will be performed to assess a vascular etiology before the treatment and 2 weeks later. The patients will be randomized into a treatment group (12 patients) and a control group (12 patients).

All patients will sign an informed consent. The treatment group will be injected IC with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) for color Doppler assessment, followed, next day by 50 units of BTX-A. The control group, 12 patients, will be injected with the trimix solution during penile color Doppler assessment followed next day with a normal saline injection. The erection hardness score (EHS) will be assessed during the Doppler exam.

Procedure: At least 1 day after the penile color Doppler test, the patient is placed in the supine position flaccid and stretched penile length and girth would be measured from tip of the penis to the pubic bone will be done. A rubber band will be applied to the base of the penis. The skin will be prepped with alcohol swabs followed by the IC injection of 50 units of BTX-A. Direct pressure will be applied for 2 minutes. The rubber band will be removed after 15 minutes.

Patients and controls will fill the Sexual Health Inventory for men (SHIM) questionnaire and answer the the Sexual Encounter Profile questions 1 and 2 (SEP 2 & SEP 3), and the global assessment question (GAQ) before and 4 weeks after treatment.

The rational for selecting the minimum 2-weeks waiting period is to give a chance for the BTX-A to reach its maximum effect. Possible Risks include pain and prolonged erections.

ELIGIBILITY:
Inclusion Criteria:

* 24 males will be included in the study recruited from Andrology, Sexology & STD's outpatient clinic, Kasr El Aini Hospitals, Cairo University, complaining of Vascular ED proved by penile duplex.
* Unable to develop erections sufficient for intercourse.
* Failing to respond to first line and second line treatments for Erectile Dysfunction with surgery as the only remaining treatment option.
* Age between 40 to 70 years.

Exclusion Criteria:

* Significant cardiovascular disease interfering with sexual activity

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Ghanem, MD, FECSM, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Cairo Governorate, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started Nov 1, 2015 Completed May 24, 2016 Cairo University Andrology outpatient clinic
Groups:
- Study Group: The treatment group, 12 patients will be injected intracavernously with a trimix solution for colour Doppler assessment, followed, on a separate day by 50 units of Botulinum toxin (BTX) A.
  Botulinum Toxin Type A: The treatment group will be injected intracavernously with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) for colour Doppler assessment, followed next day by 50 units of BTX-A.
- Control Group: The control group, 12 patients, will be injected with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) during penile colour Doppler assessment followed on a separate day with a normal saline injection.
  Normal Saline: The control group, 12 patients, will be injected with a trimix solution during penile colour Doppler assessment followed next day with a normal saline injection.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (BTX) A Group | Saline Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 52.1 [40 to 66] | 55.1 [51 to 62] | 53.6 [40 to 66]
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Egypt | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cavernosal Artery Mean PSV Before Treatment
Description: Baseline mean Peak systolic velocity (PSV) in the Cavernosal arteries, on color Doppler examination, in the patient and control groups, before treatment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- (BTX) A: The treatment group will be injected intracavernously with a trimix solution for colour Doppler assessment, followed, on a separate day by 50 units of Botulinum toxin (BTX) A.
  Botulinum Toxin Type A: The treatment group will be injected intracavernously with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) for colour Doppler assessment, followed next day by 50 units of BTX-A.
Arm/Group | (BTX) A | Saline Group
Number analyzed (Participants) | 12 | 12
cm/s | 24.5 (4.80) | 28.2 (9.79)

2. Primary Outcome: Cavernosal Artery Mean PSV After Treatment
Description: Cavernosal artery mean peak systolic velocity (PSV) after treatment, on color Doppler examination, in the patient and control groups.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
cm/s | 34.0 (9.32) | 30.5 (16.4)
Statistical Analysis 1: Comparison: (BTX) A Group; Comparing the mean PSV before & after treatment in the study group using the t-test; Test type: Superiority or Other; p = 0.0049, t-test, 1 sided
Statistical Analysis 2: Comparison: Saline Group; Comparing the mean PSV before & after treatment in the control group using the t-test; Test type: Superiority or Other; p = 0.68, t-test, 1 sided

3. Secondary Outcome: EHS Before Treatment
Description: Clinical assessment of the Erection hardness score (EHS) in both groups after ICI at baseline.
  The Erection Hardness Score (EHS) is designed to measure the rigidity of erection. It ranges from 0 (no erection) to 4 (Fully rigid and hard erection).
  0 - Penis does not enlarge.
  1. - Penis is larger, but not hard.
  2. - Penis is hard, but not hard enough for penetration.
  3. - Penis is hard enough for penetration, but not completely hard.
  4. - Penis is completely hard and fully rigid. The average score is reported for each group.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on EHS scale
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
units on EHS scale | 2.08 (0.515) | 2.17 (0.577)

4. Secondary Outcome: EHS After Treatment
Description: Clinical assessment of the Erection hardness score (EHS) in both groups after ICI after 2 weeks.
  The Erection Hardness Score (EHS) is designed to measure the rigidity of erection. It ranges from 0 (no erection) to 4 (Fully rigid and hard erection).
  0 - Penis does not enlarge.
  1. - Penis is larger, but not hard.
  2. - Penis is hard, but not hard enough for penetration.
  3. - Penis is hard enough for penetration, but not completely hard.
  4. - Penis is completely hard and fully rigid. The average score is reported for each group.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on EHS scale
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
units on EHS scale | 2.75 (0.622) | 2.17 (0.389)
Statistical Analysis 1: Comparison: (BTX) A Group; Comparing the Erection hardness score before & after treatment in the study group; Test type: Superiority or Other; p = 0.01086956, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Saline Group; Comparing the Erection hardness score before & after treatment in the control group; Test type: Superiority or Other; p = 0.6618176, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: SHIM Score Before Treatment
Description: Assessment of the Sexual Health Inventory for men (SHIM) questionnaire before treatment for both groups. It is a questionnaire that helps asses if the patient has erectile dysfunction (ED) and assesses its degree. Results range from 1 to 25. A score of 1-7 denotes Severe ED, 8-11 Moderate ED, 12-16, Mild to Moderate ED, 17-21 Mild ED, 22-25 No ED.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on the SHIM scale
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
units on the SHIM scale | 5.58 (1.93) | 5.75 (2.30)

6. Secondary Outcome: SHIM Score After Treatment
Description: as for outcome 5
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on SHIM scale
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
units on SHIM scale | 10.3 (5.38) | 6.67 (3.68)
Statistical Analysis 1: Comparison: (BTX) A Group; SHIM Score in the study group before & after treatment; Test type: Superiority or Other; p = 0.00751288, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Saline Group; SHIM Score in the control group before & after treatment; Test type: Superiority or Other; p = 0.6618176, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Global Assessment Question (GAQ)
Description: Assessment of the effect of treatment by asking "Has the treatment you have been taking improved your erectile function?". The number answering "Yes" in both the treatment and control groups are calculated.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
participants | 7 | 1
Statistical Analysis 1: Comparison: (BTX) A Group vs Saline Group; Test type: Superiority or Other; p = 0.027191, Fisher Exact — Due to the small sample size Fisher exact test was chosen. 7 out of 12 in the treatment group answered "yes", while 1 out of 12 in the control group answered "yes"

8. Secondary Outcome: SEP-Q2 Question Before Treatment
Description: Number of patients answering "Yes" to the Sexual Encounter Profile question 2 (SEP-Q2: Were you able to insert your penis into your partner's vagina?)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
participants | 0 | 2

9. Secondary Outcome: SEP-Q2 Question After Treatment
Description: Number of patients answering "Yes" to the Sexual Encounter Profile question 2 (SEP-Q2: Were you able to insert your penis into your partner's vagina?) after treatment.
  This analysis compares the number of patients who were able to perform vaginal intromission (insert the penis into the partner's vagina) after treatment in the (BTX) A group versus the Saline group.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
participants | 7 | 2
Statistical Analysis 1: Comparison: (BTX) A Group vs Saline Group; Fisher Exact Test was used to compare the change in the number of in patients who answered "Yes" in Secondary Outcome 8 (SEP-Q2 Question Before Treatment) to patients who answered "Yes" in Secondary Outcome 9 (SEP-Q2 Question after Treatment), for both (BTXA) and Saline groups; Test type: Superiority or Other; p = 0.109091, Fisher Exact

10. Secondary Outcome: SEP-Q3 Question Before Treatment
Description: Number of patients answering "Yes" to the Sexual Encounter Profile question 3 (SEP-Q3: Did your erection last long enough for you to have successful intercourse?) before treatment.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

11. Secondary Outcome: SEP-Q3 Question After Treatment
Description: Number of patients answering "Yes" to the Sexual Encounter Profile question 3 (SEP-Q3: Did your erection last long enough for you to have successful intercourse?) after treatment.
  This analysis compares the number of patients who were able to maintain their erection long enough to complete sexual intercourse after treatment in the (BTX) A group versus the Saline group.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | (BTX) A Group | Saline Group
Number analyzed (Participants) | 12 | 12
participants | 3 | 1
Statistical Analysis 1: Comparison: (BTX) A Group vs Saline Group; Fisher Exact Test was used to compare the change in patients who answered "Yes" in Secondary Outcome 10 (SEP-Q3 Question Before Treatment) to patients who answered "Yes" in Secondary Outcome 11 (SEP-Q3 Question after Treatment); Test type: Superiority or Other; p = 1, Fisher Exact

ADVERSE EVENTS:
Arm/Group | (BTX) A Group | Saline Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Small sample size (24 total). Several questions need answering: Would a higher BTX-A give a better result? Would the results be maintained for the expected duration of BTX-A effectiveness period of 3 to 6 months?

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes